CLINICAL TRIAL: NCT07372300
Title: The Efficacy of Combination of Modulated Electro-Hyperthermia(mEHT) in The Multimodality Management in Locally Advanced Rectal Cancer: A Multicenter Phase 3 Randomized Control Trial.
Brief Title: Modulated Electro-Hyperthermia in Combination With Multimodal Therapy for Locally Advanced Rectal Cancer
Acronym: mEHT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shih-Kai Hung (Other)
Collaborators: Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Shih-Kai Hung, Director of Radiation Oncology, Dalin Tzu Chi General Hospital
Organization: Dalin Tzu Chi General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iIRB No. A11304001; iIRB No. A11304001 (Other: Dalin Tzu Chi Hospital - Research Ethics Committee)
Record Dates: First submitted 2026-01-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Rectal Carcinoma
Keywords: Rectal cancer; Hyperthermia; Neoadjuvant; Radiotherapy; Downstaging
MeSH Terms: conditions — Rectal Neoplasms; Hyperthermia | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNT + mEHT (Experimental): Participants receive standard TNT with modulated electro-hyperthermia (mEHT). This includes long-course CRT with concurrent mEHT, twice weekly, for 5-6 weeks, followed by neoadjuvant chemotherapy (4-6 months), and finally surgery.
  Chemoradiation therapy phase Drug: Capecitabine or Tegafur/ Uracil or Fluorouracil (5-FU) + Leucrorin (LV) concomitant with RT Procedure: Radiotherapy Total radiation dose of 45-50.4 Gy delivered in 25-28 fractions to the pelvis, and the dose of 52-56 Gy for gross tumor volumes and positive lymph nodes.
  Device: Oncotherm Modulated EHY-2030 Oncotherm device is working on a radiofrequency of 13.56 MHz. Treatments are administered twice weekly during the 5-6-week CRT phase. Each session lasts 60 minutes
  Neoadjuvant systemic therapy:
  4-6 months of neoadjuvant chemotherapy using CAPEOX or mFOLFOX 6 regimens following CRT
  Surgery:
  Total mesorectal excision (TME) performed after the completion of neoadjuvant chemotherapy.
  Interventions: Device: Hyperthermia
- TNT alone (No Intervention): Participants receive standard TNT without modulated electro-hyperthermia (mEHT).
  This includes long-course CRT with concurrent mEHT, twice weekly, for 5-6 weeks, followed by neoadjuvant chemotherapy (4-6 months), and finally surgery.
  Chemoradiation therapy phase Drug: Capecitabine or Tegafur/ Uracil or Fluorouracil (5-FU) + Leucrorin (LV) concomitant with RT Procedure: Radiotherapy Total radiation dose of 45-50.4 Gy delivered in 25-28 fractions to the pelvis, and the dose of 52-56 Gy for gross tumor volumes and positive lymph nodes.
  Device: Oncotherm Modulated EHY-2030
  Neoadjuvant systemic therapy:
  4-6 months of neoadjuvant chemotherapy using CAPEOX or mFOLFOX 6 regimens following CRT
  Surgery:
  Total mesorectal excision (TME) performed after the completion of neoadjuvant chemotherapy.

INTERVENTIONS:
Device: Hyperthermia — Modulated electro-hyperthermia, 2 times weekly for 6 weeks
  Arms: TNT + mEHT

SUMMARY:
The goal of this clinical trial is to investigate if the addition of modulated electro-hyperthermia (mEHT) improves tumor down-staging and pathological response in adult patients (20 years and above) with locally advanced rectal adenocarcinoma (cT3N0M0 with high risk of recurrence, cT3N1-2M0, or cT4N0-2M0). The main questions it aims to answer are:

* Does the addition of mEHT to the Total Neoadjuvant Therapy (TNT) regimen significantly increase the rate of tumor down-staging (ypT and ypN) compared to TNT alone?
* Does the combination therapy improve the pathological complete response (pCR) rate and long-term outcomes (such as disease-free survival) compared to standard TNT?

Researchers will compare participants randomized to receive Total Neoadjuvant Therapy (TNT) plus mEHT using the Oncotherm EHY-2030 device to participants receiving TNT alone to see if the adjunctive mEHT therapy enhances tumor regression and improves patient prognosis. Participants will be randomized (1:1) into one of the two groups and will undergo the following regimen:

* Receive standard TNT, which includes 5-6 weeks of chemoradiotherapy (CRT) followed by 4-6 months of neoadjuvant chemotherapy.
* Patients in the experimental group will receive mEHT twice a week during the CRT period.

DETAILED DESCRIPTION:
This study is designed as a pivotal Phase 3, open-label, two-treatment group, multi-institute randomized control trial (1:1).

Study Population & Allocation:

Participants with pathologically confirmed rectal adenocarcinoma who are recommended for TNT by a specialist surgeon will be included. Patients are randomly allocated (1:1) into either the Experimental Arm (TNT + mEHT combination) or the Control Arm (TNT alone).

Intervention and Device:

Modulated electro-hyperthermia (mEHT, trade name Oncotherm) will be delivered using the Oncotherm EHY-2030 device. This technique uses electromagnetic waves at 13.56 MHz and incorporates a low-frequency current wave to deliver energy selectively to the cancerous area. The Oncotherm computer system automatically adjusts the optimal frequency, introducing random resonance to heat the tumor tissue and improve the tumor microenvironment. Local hyperthermia is intended to control tumors by raising the local body temperature to 39℃-42℃.

We hypothesized that the combination of hyperthermia with other treatments (such as radiotherapy and chemotherapy) can improve treatment outcome without additional toxicity. Patients in the Experimental Arm will receive mEHT twice a week specifically during the CRT period.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 years and above
2. Gender: Not restricted
3. Initial pathological diagnosis of adenocarcinoma of the rectum
4. Expected survival ≥ six months
5. Clinical staging of cT3N0 with high recurrence risk or cT3N1-2 or cT4N0-2 rectal cancer, requiring neoadjuvant therapy, without distant metastasis; must meet the following tumor definitions [staging system according to the 8th edition of the AJCC staging manual]:

   1. cT3: Tumor invades through the muscularis propria into pericolorectal tissues
   2. cT4a: Tumor invades through the visceral peritoneum (including gross perforation of the bowel through tumor and continuous invasion of tumor through areas of inflammation to the surface of the visceral peritoneum)
   3. cT4b: Tumor directly invades or adheres to adjacent organs or structures *High recurrence risk factors: cT3 tumor ≤ 5 cm from the anal verge or MRI showing circumferential resection margin (CRM) < 0.2 cm; cT4 tumor or cN2, presence of MRI showing extramural vascular invasion.

7. ECOG performance status: 0 - 2 8. Healthy condition suitable for standard treatment, including 25 to 30 fractions of long-course radiotherapy and concurrent chemotherapy (capecitabine or fluorouracil) and subsequent 4- to 6-month chemotherapy, including modified FOLFOX-6 or CAPEOX 9. Willingness to participate in the clinical trial and signed the informed consent form for the protocol.

Exclusion Criteria:

* (e) Active infection or severe underlying disease making the patient unsuitable for the trial treatments
* Known HIV infection
* Untreated thyroid disease
* Active Crohn's disease or ulcerative colitis
* Other systemic autoimmune diseases 9. History of any physical or mental disorder resulting the patient unable to understand or comply with trial requirements, or diminished social communication ability, or unable to provide informed consent 10. Known allergic reaction to trial medications 11. Pregnant or breastfeeding women 12. Substance or alcohol dependence within six months before screening 13. Inability to comply with treatment, assessments, or follow-up

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Down-staging Rate | Time Frame: 9 months from the date of randomization
  Evaluation of the decrease in ypT and ypN staging for patients with locally advanced rectal cancer following the current recommended treatment method, total neoadjuvant therapy (TNT). The ycT and ycN staging will be assessed using MRI within three months post-treatment for patients who do not undergo surgery.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate. | 9 months from the date of randomization
  A pCR must include no gross or microscopic tumor identified anywhere within the surgical specimen. This must include:
  * No evidence of malignant cells in the primary tumor specimen AND
  * No evidence of malignant cells in the lymph nodes.
Treatment Response Patterns | 9 months
  Using the Dworak Scale, defined as "good tumor shrinkage" with Grade 3 and Grade 4.
Overall Survival (OS) | 12, 36, 60 months from the date of randomization
  OS is defined as time from randomization to the date of death due to any cause.
Disease-Free Survival (DFS) | 12, 36, 60 months from the date of randomization
  DFS is defined as the time from randomization to the date of local recurrence, regional recurrence, distant recurrence or death due to all causes whichever comes first. Patients who fail to return for evaluation after beginning therapy will be censored for DFS on the last day of therapy.
Local Control Rate (LCR) | Time Frame: 12, 36, 60 months from the date of randomization.
  LCR is defined as the time from randomization to the date of the first documentation of local recurrence.
Distant Metastasis-Free Survival (DMFS) | 12, 36, 60 months from the date of randomization
  DMFS is defined as the time from randomization to the date of the first documentation of distant metastasis.
Colostomy-Free Survival (CFS) | 12, 36, 60 months from the date of randomization.
  CFS is defined as being alive without a colostomy, excluding colostomies reversed during follow-up.
Comparison of Surgery Rates | 12 months
  Comparison of Surgery Rates is defined as the rate of patients who receive TME between two groups after TNT.
Surgical Techniques | 12 months
  Surgical Techniques to be recorded: Total Mesorectal Excision (TME), local excision or other (specify).
Number of Hyperhermia | 9 months
  For the optimal treatment, patients in experimental arm receive hyperthermia by using Oncotherm EHY-2030 device, with a planned power output of 60 minutes. The number of treatment where this optimal output could not be reached must be recorded and reported.
Adverse Effects Assessment | 2, 36, 60 months
  Using CTCAE v5.0, scored 0 - 5, with higher scores indicating more severe adverse effects. The items include: radiation dermatitis, anorexia, nausea, vomiting, constipation, diarrhea, dysuria, hematuria, and fatigue. All items are planned to be evaluated at the initiation of treatment (week 1), and subsequently at the week 6, week 9, week 28, week 42, week 48, week 60, week 72, week 84, and week 96 (+/- 3 weeks is permitted).
The effect of treatment on white blood cell count | 2, 36, 60 months
  Recording total white cell counts, absolute neutrophil counts, and absolute lymphocyte counts of all patients. Blood samples are obtained at the initiation of treatment (week 1), and subsequently at the week 6, week 9, week 28, week 42, week 48, week 60, week 72, week 84, and week 96 (+/- 3 weeks is permitted).
The effect of treatment on hemoglobin level | 2, 36, 60 months
  Recording hemoglobin levels of all patients. Blood samples are obtained at the initiation of treatment (week 1), and subsequently at the week 6, week 9, week 28, week 42, week 48, week 60, week 72, week 84, and week 96 (+/- 3 weeks is permitted).
The effect of treatment on platelet count | 2, 36, 60 months
  Recording platelet counts of all patients. Blood samples are obtained at the initiation of treatment (week 1), and subsequently at the week 6, week 9, week 28, week 42, week 48, week 60, week 72, week 84, and week 96 (+/- 3 weeks is permitted).
Late Radiation Therapy Adverse Effects | 36, 60 months
  Using the LENT/SOMA scoring system, evaluating symptoms such as tenesmus, mucosal loss, sphincter control, stool frequency, pain, bleeding, ulceration, stricture, etc., scored 1 - 4, with higher scores indicating worse outcomes.
Quality of Life Analysis | 12 months.
  Quality of Life (QoL) assessment is mandatory for all eligible patients randomized into the trial. QoL will be evaluated using the total score of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). A printed questionnaire will be administered in the clinic by a CRA or study nurse at the following time points:
  * Baseline (at the time of randomization, prior to treatment initiation).
  * The last week of neoadjuvant CRT with or without mEHT.
  * Nine months after the completion of the TNT course (approximately 42 weeks ± 3 weeks post-randomization).
Rectal Cancer Quality of Life Analysis | 12 months.
  Rectal Cancer Quality of Life (QoL) assessment is mandatory for all eligible patients randomized into the trial. QoL will be evaluated using the total score of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-CR29). A printed questionnaire will be administered in the clinic by a CRA or study nurse at the following time points:
  * Baseline (at the time of randomization, prior to treatment initiation).
  * The last week of neoadjuvant CRT with or without mEHT.
  * Nine months after the completion of the TNT course (approximately 42 weeks ± 3 weeks post-randomization).
Functional Assessment Post Rectal Cancer Surgery | 12 months
  Using the LAR score.
  The QoL evaluation focus on functional outcome will be evaluated using LAR score. This assessment is mandatory for all eligible patients randomized into the trial. A printed questionnaire will be administered in the clinic by a CRA or study nurse at the following time points:
  * Baseline (at the time of randomization, prior to treatment initiation).
  * The last week of neoadjuvant CRT with or without mEHT.
  * Nine months after the completion of the TNT course (approximately 42 weeks ± 3 weeks post-randomization).

CONTACTS AND LOCATIONS:
Locations (1):
- Dalin Tzu Chi Hospital, Chiayi City, Dalin Township, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Aguilar J, Patil S, Gollub MJ, Kim JK, Yuval JB, Thompson HM, Verheij FS, Omer DM, Lee M, Dunne RF, Marcet J, Cataldo P, Polite B, Herzig DO, Liska D, Oommen S, Friel CM, Ternent C, Coveler AL, Hunt S, Gregory A, Varma MG, Bello BL, Carmichael JC, Krauss J, Gleisner A, Paty PB, Weiser MR, Nash GM, Pappou E, Guillem JG, Temple L, Wei IH, Widmar M, Lin S, Segal NH, Cercek A, Yaeger R, Smith JJ, Goodman KA, Wu AJ, Saltz LB. Organ Preservation in Patients With Rectal Adenocarcinoma Treated With Total Neoadjuvant Therapy. J Clin Oncol. 2022 Aug 10;40(23):2546-2556. doi: 10.1200/JCO.22.00032. Epub 2022 Apr 28. PMID 35483010
- [Background] Park JH, Yoon SM, Yu CS, Kim JH, Kim TW, Kim JC. Randomized phase 3 trial comparing preoperative and postoperative chemoradiotherapy with capecitabine for locally advanced rectal cancer. Cancer. 2011 Aug 15;117(16):3703-12. doi: 10.1002/cncr.25943. Epub 2011 Feb 15. PMID 21328328
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] Shen MH, Chen LP, Ho TF, Shih YY, Huang CS, Chie WC, Huang CC. Validation of the Taiwan Chinese version of the EORTC QLQ-CR29 to assess quality of life in colorectal cancer patients. BMC Cancer. 2018 Apr 2;18(1):353. doi: 10.1186/s12885-018-4312-y. PMID 29606101
- [Background] Rubin P, Constine LS, Fajardo LF, Phillips TL, Wasserman TH. RTOG Late Effects Working Group. Overview. Late Effects of Normal Tissues (LENT) scoring system. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1041-2. doi: 10.1016/0360-3016(95)00057-6. No abstract available. PMID 7713774
- [Background] Dworak O, Keilholz L, Hoffmann A. Pathological features of rectal cancer after preoperative radiochemotherapy. Int J Colorectal Dis. 1997;12(1):19-23. doi: 10.1007/s003840050072. PMID 9112145
- [Background] De Haas-Kock DF, Buijsen J, Pijls-Johannesma M, Lutgens L, Lammering G, van Mastrigt GA, De Ruysscher DK, Lambin P, van der Zee J. Concomitant hyperthermia and radiation therapy for treating locally advanced rectal cancer. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD006269. doi: 10.1002/14651858.CD006269.pub2. PMID 19588384
- [Background] Liu S, Jiang T, Xiao L, Yang S, Liu Q, Gao Y, Chen G, Xiao W. Total Neoadjuvant Therapy (TNT) versus Standard Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer: A Systematic Review and Meta-Analysis. Oncologist. 2021 Sep;26(9):e1555-e1566. doi: 10.1002/onco.13824. Epub 2021 Jun 7. PMID 33987952
- [Background] Conroy T, Bosset JF, Etienne PL, Rio E, Francois E, Mesgouez-Nebout N, Vendrely V, Artignan X, Bouche O, Gargot D, Boige V, Bonichon-Lamichhane N, Louvet C, Morand C, de la Fouchardiere C, Lamfichekh N, Juzyna B, Jouffroy-Zeller C, Rullier E, Marchal F, Gourgou S, Castan F, Borg C; Unicancer Gastrointestinal Group and Partenariat de Recherche en Oncologie Digestive (PRODIGE) Group. Neoadjuvant chemotherapy with FOLFIRINOX and preoperative chemoradiotherapy for patients with locally advanced rectal cancer (UNICANCER-PRODIGE 23): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 May;22(5):702-715. doi: 10.1016/S1470-2045(21)00079-6. Epub 2021 Apr 13. PMID 33862000
- [Background] Jin J, Tang Y, Hu C, Jiang LM, Jiang J, Li N, Liu WY, Chen SL, Li S, Lu NN, Cai Y, Li YH, Zhu Y, Cheng GH, Zhang HY, Wang X, Zhu SY, Wang J, Li GF, Yang JL, Zhang K, Chi Y, Yang L, Zhou HT, Zhou AP, Zou SM, Fang H, Wang SL, Zhang HZ, Wang XS, Wei LC, Wang WL, Liu SX, Gao YH, Li YX. Multicenter, Randomized, Phase III Trial of Short-Term Radiotherapy Plus Chemotherapy Versus Long-Term Chemoradiotherapy in Locally Advanced Rectal Cancer (STELLAR). J Clin Oncol. 2022 May 20;40(15):1681-1692. doi: 10.1200/JCO.21.01667. Epub 2022 Mar 9. PMID 35263150
- [Background] Dijkstra EA, Nilsson PJ, Hospers GAP, Bahadoer RR, Meershoek-Klein Kranenbarg E, Roodvoets AGH, Putter H, Berglund A, Cervantes A, Crolla RMPH, Hendriks MP, Capdevila J, Edhemovic I, Marijnen CAM, van de Velde CJH, Glimelius B, van Etten B; Collaborative Investigators. Locoregional Failure During and After Short-course Radiotherapy Followed by Chemotherapy and Surgery Compared With Long-course Chemoradiotherapy and Surgery: A 5-Year Follow-up of the RAPIDO Trial. Ann Surg. 2023 Oct 1;278(4):e766-e772. doi: 10.1097/SLA.0000000000005799. Epub 2023 Jan 20. PMID 36661037
- [Background] Bahadoer RR, Dijkstra EA, van Etten B, Marijnen CAM, Putter H, Kranenbarg EM, Roodvoets AGH, Nagtegaal ID, Beets-Tan RGH, Blomqvist LK, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes A, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; RAPIDO collaborative investigators. Short-course radiotherapy followed by chemotherapy before total mesorectal excision (TME) versus preoperative chemoradiotherapy, TME, and optional adjuvant chemotherapy in locally advanced rectal cancer (RAPIDO): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):29-42. doi: 10.1016/S1470-2045(20)30555-6. Epub 2020 Dec 7. PMID 33301740
- [Background] Dewdney A, Cunningham D, Tabernero J, Capdevila J, Glimelius B, Cervantes A, Tait D, Brown G, Wotherspoon A, Gonzalez de Castro D, Chua YJ, Wong R, Barbachano Y, Oates J, Chau I. Multicenter randomized phase II clinical trial comparing neoadjuvant oxaliplatin, capecitabine, and preoperative radiotherapy with or without cetuximab followed by total mesorectal excision in patients with high-risk rectal cancer (EXPERT-C). J Clin Oncol. 2012 May 10;30(14):1620-7. doi: 10.1200/JCO.2011.39.6036. Epub 2012 Apr 2. PMID 22473163
- [Background] Ma B, Gao P, Wang H, Xu Q, Song Y, Huang X, Sun J, Zhao J, Luo J, Sun Y, Wang Z. What has preoperative radio(chemo)therapy brought to localized rectal cancer patients in terms of perioperative and long-term outcomes over the past decades? A systematic review and meta-analysis based on 41,121 patients. Int J Cancer. 2017 Sep 1;141(5):1052-1065. doi: 10.1002/ijc.30805. Epub 2017 Jun 8. PMID 28560805
- [Background] Roh MS, Colangelo LH, O'Connell MJ, Yothers G, Deutsch M, Allegra CJ, Kahlenberg MS, Baez-Diaz L, Ursiny CS, Petrelli NJ, Wolmark N. Preoperative multimodality therapy improves disease-free survival in patients with carcinoma of the rectum: NSABP R-03. J Clin Oncol. 2009 Nov 1;27(31):5124-30. doi: 10.1200/JCO.2009.22.0467. Epub 2009 Sep 21. PMID 19770376
- [Background] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Background] Wo JY, Anker CJ, Ashman JB, Bhadkamkar NA, Bradfield L, Chang DT, Dorth J, Garcia-Aguilar J, Goff D, Jacqmin D, Kelly P, Newman NB, Olsen J, Raldow AC, Ruiz-Garcia E, Stitzenberg KB, Thomas CR Jr, Wu QJ, Das P. Radiation Therapy for Rectal Cancer: Executive Summary of an ASTRO Clinical Practice Guideline. Pract Radiat Oncol. 2021 Jan-Feb;11(1):13-25. doi: 10.1016/j.prro.2020.08.004. Epub 2020 Oct 21. PMID 33097436
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- See also: Network NCC. Rectal Cancer (Version 2.2024). — https://www.nccn.org/professionals/physician_gls/pdf/rectal.pdf